CLINICAL TRIAL: NCT05669118
Title: Dental Autotransplantation or Immediate Single Implant for the Replacement of a Hopeless Molar: a Comparative Case Series Study.
Brief Title: Dental Autotransplantation or Immediate Single Implant for the Replacement of a Hopeless Molar.
Status: Completed | Type: Observational
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, Principal Investigator, Aula Dental Avanzada
Other Study IDs: PROSP AUTO
Record Dates: First submitted 2022-12-08; First posted 2022-12-30 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Transplantation, Autologous; Autografts; Surgery, Oral
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autotransplantation: Patients who receive one tooth autotransplanted.
  Interventions: Procedure: Tooth Autotransplantation
- Immediate implant: Patients who receive one inmediate dental implant.
  Interventions: Procedure: Immediate implant

INTERVENTIONS:
Procedure: Tooth Autotransplantation — Place another tooth in the place of the newly extracted tooth in the same patient.
  Other Names: Dental autotransplant
  Groups: Autotransplantation
Procedure: Immediate implant — Place a dental implant immediately after tooth extraction.
  Other Names: Type 1 implant
  Groups: Immediate implant

SUMMARY:
The aim of this comparative study is to know the differences between the soft tissue volume changes around the autotransplanted tooth and the dental implant placed immediately after the extraction of a posterior tooth. Patient-centered results will also be obtained after having received one or the other treatment.

DETAILED DESCRIPTION:
Dental autotransplantation has high levels of success in permanent teeth with open apex. The results of success in permanent teeth with closed apex are somewhat lower but sufficient to consider the treatment as a viable alternative and to extend the therapeutic range of the treatment to older ages.

The aim of this prospective observational investigation is to evaluate the dimensional and attachment changes that occur in the treated areas and in the autotransplanted teeth respectively of adult patients with permanent teeth with closed apex. All adult patients receiving a dental autotransplantation between the years 2022 and 2023 will be included.

Pre-treatment, volume and insertion parameters will be recorded before and one year after treatment. The comparison with the extraction and dental implant treatment will be made using the digital records that are usually obtained during the performance of this treatment. The comparison will be made with the same number of patients who have been recruited for the dental autotransplant treatment, and the volumetric changes that occur will also be analyzed.

The volume comparisons will be carried out using the Medit Link digital measurement software (Medit, Seoul, Republic of Korea) and data will be obtained and analyzed statistically in order to draw the appropriate conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Patients in ASA-I health status
* Aged between 18 and 80 years,
* Present a tooth in need of extraction with a mature candidate donor tooth compatible with the recipient bed
* Acceptance of proposed treatment of dental autotransplantation

Exclusion Criteria:

* Unavailability of a candidate donor tooth
* Refusal of proposed treatment of dental autotransplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who come to the clinic and need a tooth extracted.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Soft tissue volume changes | 2 times measurement: day 0 and 6 months after
  Soft tissue volume changes in the buccal side of the site in mm3
Periodontal probing pocket depth | 6 months after
  Periodontal probing pocket depth in mm

SECONDARY OUTCOMES:
Patients satisfaction after treatment | 6 months after the reception of the treatment
  Satisfaction assessed by Numeric Rating Scale (NRS) form 0 to 10, being 0 "not satisfied at all" and 10 "very satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Esteve-Pardo, PhD, Principal Investigator — Clínica Dental Esteve
Locations (1):
- Clínica Dental Esteve, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request.